CLINICAL TRIAL: NCT03291912
Title: Therapeutic Effect of Adjuvant Chuna Manual Therapy (CMT) in Subjects With Cervicogenic Dizziness: a Prospective, Pragmatic, Assessor-blind, Randomized Controlled Trial
Brief Title: Chuna Manual Therapy for Cervicogenic Dizziness
Acronym: CHERIE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This registration has moved to a local ICTRP (CRIS; https://cris.nih.go.kr, KCT0002565).
Sponsor: Kyunghee University (Other)
Responsible Party: Principal Investigator, Lee Eui-ju, Professor, Ph.D. KMD., Kyunghee University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HB16C0010-CMT
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Cervicogenic Dizziness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chuna Manual Therapy (CMT) (Experimental): 1. Chuna manual therapy (CMT), 2 sessions/week, 6 weeks (12 sessions in total)
  2. Usual care therapy (UC), 2 sessions/week, 6 weeks (12 sessions in total)
     * Usual care consists of physical therapy and patients education. Physical therapy consists of meridian muscle interferential current electricity (or meridian transcutaneous electricity) and hot pack (or infrared lamp).
     * Patients will be educated about cause and risk factors of cervicogenic dizziness, general neck muscle functions, self-exercising for relieving the symptoms.
     * CMT and UC group will receive the same UC regimen.
  Interventions: Procedure: Chuna Manual Therapy; Procedure: Usual care
- Usual Care (UC) (Active Comparator): Usual care therapy (UC), 2 sessions/week, 6 weeks (12 sessions in total)
  * Usual care consists of physical therapy and patients education. Physical therapy consists of meridian muscle interferential current electricity (or meridian transcutaneous electricity) and hot pack (or infrared lamp).
  * Patients will be educated about cause and risk factors of cervicogenic dizziness, general neck muscle functions, self-exercising for relieving the symptoms.
  * CMT and UC group will receive the same UC regimen.
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Chuna Manual Therapy — * Unique manual therapy in traditional Korean medicine
  * Mandatory techniques for neck part and selective techniques for other part (if necessary)
  * Selective techniques depends on a patient's condition (judged by traditional Korean medicine doctor)
  Arms: Chuna Manual Therapy (CMT)
Procedure: Usual care — 1. Physical therapy based on traditional Korean medicine theory
     * Electrical stimulation: either Meridian muscle interferential current electricity or Meridian transcutaneous electricity
     * Heat stimulation: either Hot pack or Infrared lamp
  2. Patient education
     * Physical and pathological explanation of cervicogenic dizziness
     * Cause and risk factors of cervicogenic dizziness
     * Functions of muscles related to cervicogenic dizziness
     * Home exercising to self-manage cervicogenic dizziness

SUMMARY:
This is a prospective, pragmatic, assessor-blind, randomized controlled trial to explore the effectiveness of an adjuvant Chuna manual therapy (CMT) for cervicogenic dizziness of Dizziness Handicap Inventory (DHI) ≥ 16 at baseline. Participants will be randomized and allocated to either CMT combined with usual care (UC) group or UC group with 1:1 ratio. They will receive 12 sessions of CMT or UC treatment for 6 weeks. UC consists of physical therapy and patients education.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged between 20 and 70
* neck pain and/or stiffness with dizziness, which is related to movement or positioning of cervical spine
* recurring symptom of dizziness over 1 month or more
* Dizziness Handicap Inventory ≥ 16 at baseline
* Informed consent

Exclusion Criteria:

* dizziness induced by vestibular disorders (e.g., benign paroxysmal positional vertigo, peripheral vestibulopathy, Meniere disease, vestibular neuronitis)
* dizziness induced by central nervous system (CNS) disorders (e.g., cerebellar ataxia,cerebellum infarction/hemorrhage, demyelination, vertebrobasilar insufficiency, seizure, increased intracranial pressure, Parkinson's disease, migraines)
* dizziness induced by cardiovascular disorders (e.g., arrhythmia, heart valvular disease, anemia, orthostatic hypotension, coronary artery disease)
* dizziness induced by active or uncontrolled disease (e.g., uncontrolled diabetes mellitus, hypertension, respiratory or endocrinological disorders)
* dizziness induced by side effects of medications
* severe chronic or terminal diseases (malignant cancer, tuberculosis, etc.)
* chronic psychiatric diseases under treatment (epilepsy, depression, panic disorder, etc.)
* conditions where CMT are forbidden (spinal tumor, acute fracture, infectious spondylopathy, congenital malformations of spine, operation history of spine within 3 months, progressive neurological damage, severe neurological symptoms, spinal fixation devices, syringomyelia, hydrocephaly)
* Treatment history within 1 week for cervicogenic dizziness (NSAIDs, steroid, herbal drug, acupuncture, manual therapy)
* Women of (suspected) pregnancy or breast-feeding
* Suspicion of alcohol and/or drug abuse
* Participation in another clinical study within 1 month
* Difficulty in communicating with the investigators
* Other reasons for ineligibility of participation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Dizziness Handicap Inventory (DHI) score at week 6 | Week 0, Week 6

SECONDARY OUTCOMES:
Change from baseline Dizziness Handicap Inventory (DHI) score at week 3 | Week 0, Week 3
Changes from baseline Mean Vertigo Score (MVS) at each measurement week | Week 0, Week 3, Week 6
Changes from baseline Visual Analogue Scale (VAS) score at each measurement week | Week 0, Week 3, Week 6
Changes from baseline Frequency of Dizziness score at each measurement week | Week 0, Week 3, Week 6
Changes from baseline Pain Intensity Numerical Rating Scale (PI-NRS) score at each measurement week | Week 0, Week 3, Week 6
Changes from baseline Neck Disability Index (NDI) score at each measurement week | Week 0, Week 3, Week 6
Changes from baseline Cervical Range of Motion (CROM) value at each measurement week | Week 0, Week 3, Week 6
Global Perceived Effect (GPE) score at each measurement week | Week 6
Changes from baseline Korean version of Perceived Stress Scale (K-PSS) score at each measurement week | Week 0, Week 3, Week 6
Changes from baseline EuroQoL Five Dimensions Questionnaire (EQ-5D) score at each measurement week | Week 0, Week 3, Week 6

OTHER OUTCOMES:
New Blinding Index (New BI) | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Euiju Lee, Ph.D., Principal Investigator — Kyunghee University
Locations (2):
- South Korea (2):
  - Kyung Hee University Korean Medicine Hospital, Seoul, Special Seoul City
  - Kyung Hee University Korean Medicine Hospital at Gangdong, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reid SA, Callister R, Snodgrass SJ, Katekar MG, Rivett DA. Manual therapy for cervicogenic dizziness: Long-term outcomes of a randomised trial. Man Ther. 2015 Feb;20(1):148-56. doi: 10.1016/j.math.2014.08.003. Epub 2014 Aug 27. PMID 25220110
- [Background] Li Y, Peng B. Pathogenesis, Diagnosis, and Treatment of Cervical Vertigo. Pain Physician. 2015 Jul-Aug;18(4):E583-95. PMID 26218949
- [Background] Yacovino DA, Hain TC. Clinical characteristics of cervicogenic-related dizziness and vertigo. Semin Neurol. 2013 Jul;33(3):244-55. doi: 10.1055/s-0033-1354592. Epub 2013 Sep 21. PMID 24057828
- [Background] RYAN GM, COPE S. Cervical vertigo. Lancet. 1955 Dec 31;269(6905):1355-8. doi: 10.1016/s0140-6736(55)93159-7. No abstract available. PMID 13279136
- [Background] Wrisley DM, Sparto PJ, Whitney SL, Furman JM. Cervicogenic dizziness: a review of diagnosis and treatment. J Orthop Sports Phys Ther. 2000 Dec;30(12):755-66. doi: 10.2519/jospt.2000.30.12.755. PMID 11153554
- [Background] Reid SA, Rivett DA. Manual therapy treatment of cervicogenic dizziness: a systematic review. Man Ther. 2005 Feb;10(1):4-13. doi: 10.1016/j.math.2004.03.006. PMID 15681263
- [Background] Reid SA, Rivett DA, Katekar MG, Callister R. Efficacy of manual therapy treatments for people with cervicogenic dizziness and pain: protocol of a randomised controlled trial. BMC Musculoskelet Disord. 2012 Oct 18;13:201. doi: 10.1186/1471-2474-13-201. PMID 23078200
- [Background] Karlberg M, Magnusson M, Malmstrom EM, Melander A, Moritz U. Postural and symptomatic improvement after physiotherapy in patients with dizziness of suspected cervical origin. Arch Phys Med Rehabil. 1996 Sep;77(9):874-82. doi: 10.1016/s0003-9993(96)90273-7. PMID 8822677
- [Background] Heikkila H, Johansson M, Wenngren BI. Effects of acupuncture, cervical manipulation and NSAID therapy on dizziness and impaired head repositioning of suspected cervical origin: a pilot study. Man Ther. 2000 Aug;5(3):151-7. doi: 10.1054/math.2000.0357. PMID 11034885
- [Background] Minguez-Zuazo A, Grande-Alonso M, Saiz BM, La Touche R, Lara SL. Therapeutic patient education and exercise therapy in patients with cervicogenic dizziness: a prospective case series clinical study. J Exerc Rehabil. 2016 Jun 30;12(3):216-25. doi: 10.12965/jer.1632564.282. eCollection 2016 Jun. PMID 27419118